CLINICAL TRIAL: NCT01582984
Title: Patient Understanding and Satisfaction in Informed Consent for Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: jasvinder singh (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, jasvinder singh, worker without compensation, Minneapolis Veterans Affairs Medical Center
Organization: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSPVA-124
Record Dates: First submitted 2012-04-18; First posted 2012-04-23 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Knee Arthroplasty
Keywords: consent; Patient Understanding; Knee Arthroplasty
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- iMedConsentTM and customized written handout group (Active Comparator): iMedConsentTM and a customized written handout
  Interventions: Other: video or education session in addition to standard consent
- iMedConsentTM, handout, and standard video g (Experimental): iMedConsentTM, handout, and standard AAOS video
  Interventions: Other: video or education session in addition to standard consent
- iMedConsentTM, handout, video, and formal education (Experimental): iMedConsentTM, the handout, the video, and a formal education session
  Interventions: Other: video or education session in addition to standard consent

INTERVENTIONS:
Other: video or education session in addition to standard consent — Video added to standard consent + handout Video + education session added to standard consent + handout

SUMMARY:
A structured consent process, in combination with one or a number of the aforementioned modalities (nursing education, handout, video, etc), may reasonably be expected to improve surgical informed consent. The investigators hypothesized that overall patient knowledge/retention would be influenced by the type of consent process and that more intensive training and review would result in better patient retention and recall. The investigators further hypothesized that the knowledge retention would decline following the consent process and surgery, but in a stratified manner based on the nature of preoperative teaching.

DETAILED DESCRIPTION:
please see details above

ELIGIBILITY:
Inclusion Criteria:

1. recommended total knee arthroplasty

Exclusion Criteria:

1. Unwilling to participate
2. Unable to complete questionnaire in English

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Knowledge of efficacy and complications | 6-week postoperative
  answers to questionnaire assessing knowledge

SECONDARY OUTCOMES:
knowledge regarding procedural questions with regard to the surgery and implants | Day of surgery and 6-week postoperative
  Answers to Question 4-6 on knowledge questionnaire
knowledge regarding risks of surgery | day of surgery and postoperative 6-weeks
  answers to Questions 7-9 on quetionnaire
Knowledge regarding peri- and post-operative results | day of surgery and postoperative 6-weeks
  answers to Questions 10-13 on quetionnaire
Patient satisfaction | day of surgery and postoperative 6-weeks
  answers to satisfaction Question on quetionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Terence Gioe, MD, Principal Investigator — Minneapolis VA Med crt
Locations (1):
- Minneapolis VA Medical Center, Minneapolis, Minnesota, United States